CLINICAL TRIAL: NCT00002460
Title: Phase III Randomized Study of Adjuvant Therapy With Tamoxifen vs Endocrine Ablation vs Tamoxifen Plus Endocrine Ablation vs No Adjuvant Therapy in Patients Under Age 50 With Operable Breast Cancer
Brief Title: Adjuvant Hormone Therapy in Treating Women With Operable Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CRC-PHASE-III-88002; CDR0000075539 (Registry Identifier: PDQ (Physician Data Query)); UKM-CRC-BR-UNDER 50
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2006-12

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Tamoxifen; Ovariectomy

INTERVENTIONS:
Drug: goserelin acetate
Drug: tamoxifen citrate
Procedure: ablative endocrine surgery
Procedure: oophorectomy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen.

PURPOSE: Phase III trial to compare the effectiveness of adjuvant therapy using tamoxifen or ovarian ablation with goserelin or both in treating women with stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine, in a prospective, randomized, controlled trial whether the administration of a course of adjuvant tamoxifen or ablation of ovarian function results in prolongation of time to recurrence or death in patients under 50 years of age with operable carcinoma of the breast. II. Determine how hormone manipulation affects mood and sexual functioning in these patients.

OUTLINE: This is a randomized study. Patients are stratified by clinician. All patients are randomized following primary therapy, which, in addition to surgery, may include local irradiation, perioperative cyclophosphamide, or up to 6 cycles of cyclophosphamide, methotrexate, and fluorouracil (CMF) for high-risk patients. Clinicians may elect to randomize patients to all groups or to only those groups including tamoxifen. The first group receives no further therapy. Then second group receives tamoxifen daily for at least 2 years. The third group receives ovarian ablation with goserelin via monthly injection for at least 2 years. The final group receives ovarian ablation with goserelin plus daily tamoxifen for at least 2 years. All patients are followed every 3 months for 2 years, every 6 months for 3 years, then annually.

PROJECTED ACCRUAL: 800 to 1,000 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Operable, clinical Stage I/II breast cancer (T1-3, N0-1, M0) No evidence of distant metastases on x-ray of chest, spine, and pelvis Bone scan evidence alone of secondary mass allowed unless considered unequivocal evidence of metastasis No primary carcinoma fixed to underlying muscle or chest wall No deeply fixed axillary nodes No ulceration, skin infiltration, or peau d'orange involving more than 1/3 of breast No bilateral tumors Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: Under 50 Sex: Women only Menopausal status: Any status Performance status: Not specified Life expectancy: No limits on life expectancy due to intercurrent illness Hematopoietic: WBC at least 3,000 Platelets at least 90,000 Hemoglobin at least 10 g/dL Hepatic: Normal liver function required Renal: Normal kidney function required Other: Fit for surgery No prior treatment for other malignancies except: Nonmelanomatous skin cancer Cone-biopsied in situ carcinoma of the cervix English-speaking patients eligible for quality-of-life assessments

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Chemotherapy for high-risk patients allowed at the discretion of the clinician Endocrine therapy: At least 6 weeks since prior hormonal therapy No concomitant hormonal therapy including oral contraceptives (patients must discontinue the pill for 2 years) Radiotherapy: Not specified Surgery: Not specified

Max Age: 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1987-09

CONTACTS AND LOCATIONS:
Overall Officials: Michael Baum, MD, ChM, FRCS, Study Chair — University College London Hospitals
Locations (33):
- Belgium (3):
  - Hopital De Braine-L'Alleud-Waterloo, Braine-l'Alleud
  - Institut Jules Bordet, Brussels
  - U.Z. Sint-Rafael, Leuven
- United Kingdom (30):
  - Royal Sussex County Hospital, Brighton, England
  - Castle Hill Hospital, Cottingham, England
  - Walsgrave Hospital, Coventry, England
  - Mayday University Hospital, Croydon, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Cookridge Hospital, Leeds, England
  - Whittington Hospital, London, England
  - Guy's, King's and St. Thomas' Hospitals Trust, London, England
  - Cancer Research Campaign Clinical Trials Unit-London, London, England
  - Royal Marsden NHS Trust, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - South Tees Acute Hospitals NHS Trust, Middlesbrough, Cleveland, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Derriford Hospital, Plymouth, England
  - Portsmouth Hospitals NHS Trust, Portsmouth, England
  - Salisbury General Infirmary, Salisbury, England
  - Royal South Hants Hospital, Southampton, England
  - Southampton General Hospital, Southampton, England
  - North Tees General Hospital, Stockton-on-Tees, England
  - North Staffs Royal Infirmary, Stoke-on-Trent, England
  - Radiotherapy Department, Stratford-on-Avon, Warwickshire, England
  - Sunderland Royal Infirmary, Sunderland, England
  - Royal Marsden Hospital, Sutton, England
  - Royal Hampshire County Hospital, Winchester, England
  - Belfast City Hospital Trust, Belfast, Northern Ireland
  - Mid-Ulster Hospital, Londonderry, Northern Ireland
  - Ards General Hospital, Newtownards, Northern Ireland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Velindre Hospital, Cardiff, Wales